CLINICAL TRIAL: NCT01953081
Title: A Randomized, Double-Blind Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of a Single Dose of Intravenous TD-8954 Compared With Metoclopramide in Critically Ill Patients With Enteral Feeding Intolerance
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0082
Record Dates: First submitted 2013-09-25; First posted 2013-09-30 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Enteral Feeding Intolerance
Keywords: Enteral feeding
MeSH Terms: interventions — 4-((4-((2-isopropyl-1H-benzoimidazole-4-carbonyl)amino)methyl)piperidin-1-ylmethyl)piperidine-1-carboxylic acid methyl ester; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TD-8954 (Experimental): TD-8954 single infusion for 1 hour and 4 injections of saline every 6 hours
  Interventions: Drug: TD-8954
- Metoclopramide (Active Comparator): Metoclopramide 4 doses every 6 hours for 24 hours and 1 hour infusion of saline
  Interventions: Drug: Metoclopramide

INTERVENTIONS:
Drug: TD-8954
  Arms: TD-8954
Drug: Metoclopramide
  Arms: Metoclopramide

SUMMARY:
This study is being conducted to evaluate the safety, tolerability and early efficacy of IV TD 8954 compared to metoclopramide in critically ill subjects, aged 18 to 85 years, who are admitted to the intensive care require mechanical ventilation, and are intolerant to enteral feeding.

ELIGIBILITY:
Inclusion Criteria:

* Intubated, on mechanical ventilation, and anticipated to remain on mechanical ventilation for 2 days after enrollment into the study
* Receiving enteral feeding and assessed to have developed EFI, as defined by a GRV measurement ≥250 mL within the 24 hours before randomization

Exclusion Criteria:

* History of diabetic or idiopathic gastroparesis
* Screening blood glucose >15 mmol/L (270 mg/dL) while receiving insulin
* Impaired renal function, as defined by estimated glomerular filtration rate (eGFR) <30 mL/min, as determined by the Cockcroft-Gault formula -Bilirubin concentration in blood >2 times the upper limit of normal
* ALT or AST >3 times upper limit of normal
* Alkaline phosphatase >2 times upper limit of normal
* Contraindication to enteral feeding
* Opioid or other drug overdose as the primary reason for admission to Intensive Care Unit (ICU)
* Receipt of a drug that can be used as a gastric prokinetic agent
* Receipt of agents known to directly influence the 5 HT4/acetylcholine prokinetic mechanism

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Canafax, PharmD, FCCP, Study Director — Theravance Biopharma, US, Inc.
Locations (1):
- Royal Adelaide Hospital, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chapman MJ, Jones KL, Almansa C, Barnes CN, Nguyen D, Deane AM. Blinded, Double-Dummy, Parallel-Group, Phase 2a Randomized Clinical Trial to Evaluate the Efficacy and Safety of a Highly Selective 5-Hydroxytryptamine Type 4 Receptor Agonist in Critically Ill Patients With Enteral Feeding Intolerance. JPEN J Parenter Enteral Nutr. 2021 Jan;45(1):115-124. doi: 10.1002/jpen.1732. Epub 2020 Jan 28. PMID 31990087

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TD-8954 | Metoclopramide
Started | 7 | 6
Completed | 5 | 3
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TD-8954 | Metoclopramide | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (25.29) | 55.5 (13.37) | 54.7 (19.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: the number of subjects reporting adverse events by treatment group
Time Frame: 6 Days
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | TD-8954 | Metoclopramide
Number analyzed (Participants) | 7 | 6
participants | 5 | 4

2. Primary Outcome: Gastric Retention by Scintigraphy
Description: Number of subjects with retention less than 13% at 180 minutes after dosing.
Time Frame: 180 minutes
Population: ITT
Measure: Number; unit: participants
Arm/Group | TD-8954 | Metoclopramide
Number analyzed (Participants) | 7 | 6
participants | 6 | 3

3. Secondary Outcome: Tmax
Description: Time to maximal concentration in plasma
Time Frame: 72 hours
Population: PK Analysis set for subjects receiving TD-8954, metoclopramide concentrations were not measured in the metoclopramide group.
Measure: Median (Full Range); unit: hours
Arm/Group | TD-8954 | Metoclopramide
Number analyzed (Participants) | 6 | 0
hours | 0.500 [0.500 to 1.00] |

4. Secondary Outcome: AUC
Description: Area under the plasma concentration time curve from 0 to 72 hours after dosing.
Time Frame: 72 hours
Population: One subject did not receive the full dose of TD-8954 and was excluded from PK analysis for the TD-8954 group; Metoclopramide concentrations were not measured in the Metoclopramide group.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | TD-8954 | Metoclopramide
Number analyzed (Participants) | 6 | 0
pg*hr/mL | 23200 (9240) |

5. Secondary Outcome: Cmax
Description: Maximum plasma concentration
Time Frame: 72 hours
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | TD-8954 | Metoclopramide
Number analyzed (Participants) | 6 | 0
pg/mL | 5040 (1780) |

6. Secondary Outcome: Gastric Emptying by Breath Test
Description: Time to 1/2 gastric emptying by breath test
Time Frame: 180 minutes
Population: One subject in the TD-8954 group did not receive the full dose of TD-8954 and was excluded from the TD-8954 analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | TD-8954 | Metoclopramide
Number analyzed (Participants) | 6 | 6
minutes | 135.7 (41.61) | 132.5 (53.87)

7. Secondary Outcome: Percentage Gastric Retention by Scintigraphy at 60 Minutes Postdose
Description: Mean gastric retention percentage after dosing.
Time Frame: 60 minutes
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of retention
Arm/Group | TD-8954 | Metoclopramide
Number analyzed (Participants) | 7 | 8
percentage of retention | 29.6 (36.28) | 43.3 (30.14)

8. Secondary Outcome: Percentage Gastric Retention by Scintigraphy at 120 Minutes Postdose
Description: Mean gastric retention percentage after dosing.
Time Frame: 120 minutes
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of retention
Arm/Group | TD-8954 | Metoclopramide
Number analyzed (Participants) | 7 | 8
percentage of retention | 19.6 (36.10) | 32.3 (28.32)

9. Secondary Outcome: Percentage of Gastric Retention by Scintigraphy at 240 Minutes Postdose
Description: Mean gastric retention percentage after dosing.
Time Frame: 240 minutes
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of retention
Arm/Group | TD-8954 | Metoclopramide
Number analyzed (Participants) | 7 | 8
percentage of retention | 11.1 (24.85) | 16.3 (25.64)

ADVERSE EVENTS:
Time Frame: 6 Days
Groups:
- TD-8954: TD-8954 single infusion for 1 hour and 4 injections of saline every 6 hours
  TD-8954
- Metoclopramide: Metoclopramide 4 doses every 6 hours for 24 hours and 1 hour infusion of saline
  Metoclopramide
Arm/Group | TD-8954 | Metoclopramide
Serious Adverse Events (participants affected / at risk) | 2/7 | 3/6
Other Adverse Events (participants affected / at risk) | 5/7 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TD-8954 (N=7) | Metoclopramide (N=6)
Cerebral Hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Hemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TD-8954 (N=7) | Metoclopramide (N=6)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may communicate the trial results generated by the PI, but only after the first publication or presentation of the combined study results generated by all participating sites. The Sponsor can then review trial results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days. The Sponsor cannot require changes to the communication and cannot extend the embargo.